CLINICAL TRIAL: NCT01363453
Title: Acute and Remission Therapy of Ulcerative Colitis With Oral Mesalazine
Brief Title: User Surveillance in Ulcerative Colitis
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FE999907
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Ulcerative Colitis

SUMMARY:
The aim of the non-interventional study is to document the daily doses in acute and remission therapy, the frequence of doses (1, 2, 3 or 4 times daily), when rectal dosage forms are added and, when and how long steroids are given.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to SPC
* written informed consent

Exclusion Criteria:

* contraindications according to SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private practices
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Prescription habits measured by daily dose of Mesalazine | 0 - 8 weeks

SECONDARY OUTCOMES:
Compliance measured by questionnaire for drug intake | 0 - 8 weeks
Quality of Life measured by EuroQol Questionnaire | 0 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (105):
- Germany (105):
  - Investigational , Karlsplatz 18, Aalen
  - Investigational Site, Goethestraße 5, Ansbach
  - Investigational Site, Elisenstraße 32, Aschaffenburg
  - Investigational Site, Haingasse 22, Bad Homburg
  - Investigational Site, Blankenburger Chaussee 86, Berlin
  - Investigational Site, Etkar-André-Straße 8, Berlin
  - Investigational Site, Karl-Marx-Straße 46, Berlin
  - Investigational Site, Martin-Luther-Straße 134, Berlin
  - Investigational Site, Mohrenstraße 6, Berlin
  - Investigational Site, Myslowitzer Straße 49, Berlin
  - Investigational Site, Plügerstraße 75, Berlin
  - Investigational Site, Schönhauser Allee 129, Berlin
  - Investigational Site, Hauptstraße 13 - 15, Birkenfeld
  - Investigational Site, Kurt-Schumacher-Platz 4, Bochum
  - Investigational Site, Am Burgweiher 54, Bonn
  - Investigational Site, Kasernenstraße 22 - 24, Bonn
  - Investigational Site, Münsterstraße 18, Bonn
  - Investigational Site, Trauerberg 27/28, Brandenburg
  - Investigational Site, Hermann-Hesse-Platz 3, Calw
  - Investigational Site, Moritzstraße 19, Chemnitz
  - Investigational Site, Osterstraße 44, Cloppenburg
  - Investigational Site, Leipziger Straße 45 b, Cottbus
  - Investigational Site, Münchner Straße 64, Dachau
  - Investigational Site, Schäfergraben 5 H, Delitzsch
  - Investigational Site, Hans-Böckler-Straße 20, Dinslaken
  - Investigational Site, Schadowstraße 42, Düsseldorf
  - Investigational Site, Simrockstraße 56, Düsseldorf
  - Investigational Site, Ludwig-Sandberg-Straße 4, Eberswalde
  - Investigational Site, Neuzeller Landweg 1, Eisenhüttenstadt
  - Investigational Site, Mühlendamm 23, Elmshorn
  - Investigational Site, Franz-Busbach-Str. 8, Erftstadt
  - Investigational Site, Neuwerkstraße 2, Erfurt
  - Investigational Site, Lehmanns Brink 5, Essen
  - Investigational Site, Steeler Straße 204, Essen
  - Investigational Site, Viktoriastraße 5, Euskirchen
  - Investigational Site, Sorauer Straße 56, Forst
  - Investigational Site, Im Prüfling 23, Frankfurt am Main
  - Investigational Site, Pfingstweidestraße 4, Frankfurt am Main
  - Investigational Site, Finkenstraße 31, Freising
  - Investigational Site, Bahnhofstraße 16, Fulda
  - Investigational Site, Bahnhofplatz 11, Fürth
  - Investigational Site, Straßburger Weg 4, Gelsenkirchen
  - Investigational Site, Hinter der Mauer 105, Goch
  - Investigational Site, Waldweg 1, Göttingen
  - Investigational Site, Buscheystraße 15 a, Hagen
  - Investigational Site, Drosselstraße 6 A, Hamburg
  - Investigational Site, Eppendorfer Baum 35-37, Hamburg
  - Investigational Site, Fontenay 1 d, Hamburg
  - Investigational Site, Propst-Paulsen-Straße 2, Hamburg
  - Investigational Site, Schweriner Straße 1, Hamburg
  - Investigational Site, Rathausplatz 4, Haßloch
  - Investigational Site, Kurfürstenanlage 34, Heidelberg
  - Investigational Site, Luisenstraße 18 a, Hettstedt
  - Investigational Site, Hohensachsener Str. 2, Hirschberg
  - Investigational Site, Robert-Koch-Straße 2, Hofheim
  - Investigational Site, M.-Grollmuß-Straße 10, Hoyerswerda
  - Investigational Site, J.-Lange-Straße 20, Haus 7, Jerichow
  - Investigational Site, Goethestraße 11, Kiel
  - Investigational Site, Poggendörper Weg 3-9, Kiel
  - Investigational Site, Markenbildchenweg 30, Koblenz
  - Investigational Site, Herzog-Adolph-Straße 13, Königstein im Taunus
  - Investigational Site, Schalaunische Strape 6/7, Köthen
  - Investigational Site, Friesener Straße 41, Kronach
  - Investigational Site, Auf dem Wall 6, Lindau
  - Investigational Site, Potsdamer Straße 120A, Ludwigsfelde
  - Investigational Site, Rheingönheimer Str. 121, Ludwigshafen
  - Investigational Site, Weißdornhag 2, Ludwigshafen
  - Investigational Site, Königstraße 81, Lübeck
  - Investigational Site, Pfeifferstraße 10, Magdeburg
  - Investigational Site, Weißliliengasse 31, Mainz
  - Investigational Site, Auf dem Sand 76a, Mannheim
  - Investigational Site, Zur Stadthalle 2, Merzig
  - Investigational Site, Zum Schotzberg 1 a, Merzig-Schwemmlingen
  - Investigational Site, Oldenkirchener Straße 43, Mönchengladbach
  - Investigational Site, Irisstraße 23, München
  - Investigational Site, Theodolindenstraße 97, München
  - Investigational Site, Hammer Straße 95, Münster
  - Investigational Site, Unterer Markt 26/27, Neumarkt in der Oberpfalz
  - Investigational Site, Bahnhofstraße 11, Nieder-Olm
  - Investigational Site, Glogauer Straße 42, Nuremberg
  - Investigational Site, Kleinreuther Weg 88, Nuremberg
  - Investigational Site, Weiltinger Straße 11, Nuremberg
  - Investigational Site, Hauptstraße 19, Oldenburg
  - Investigational Site, Lutherstraße 22, Oschatz
  - Investigational Site, Neue Mitte 6, Pohlheim
  - Investigational Site, Allee nach Sanssouci 7, Potsdam
  - Investigational Site, Dortustraße 4, Potsdam
  - Investigational Site, Großbeerenstraße 301, Potsdam
  - Investigational Site, R.-Breitscheid-Straße 56, Potsdam
  - Investigational Site, Hohenzollernstraße 7, Recklinghausen
  - Investigational Site, Bundesstraße 56, Roetgen
  - Investigational Site, St.-Petersburger Str. 18c, Rostock
  - Investigational Site, Heinz-Meise-Straße 101, Rotenburg (Wümme)
  - Investigational Site, Tegernseer Str. 100, Rottach-Egern
  - Investigational Site, Hoerstraße 42, Rottweil
  - Investigational Site, Neustadter Straße 61, Sonnenberg
  - Investigational Site, Winterspürer Straße 11, Stockach
  - Investigational Site, Fichteplatz 1, Strausberg
  - Investigational Site, Am Wallgraben 99, Stuttgart
  - Investigational Site, Industriestraße 4, Stuttgart
  - Investigational Site, Röhre 1, Sundern
  - Investigational Site, Olgastraße 139, Ulm
  - Investigational Site, Am Stutenteich 8, Waltrop
  - Investigational Site, Langenbeckplatz 2, Wiesbaden
  - Investigational Site, Straße von Triptis 12, Zell